CLINICAL TRIAL: NCT04617171
Title: Randomized Double Blind Placebo Controlled Trial of Benralizumab, an Antiinterleukin 5 Receptor α Monoclonal Antibody, Initiated During Hospitalization for Severe Asthma Attack in Reducing Severe Exacerbations: Phase 2B Study
Brief Title: Benralizumab Initiated During Severe Asthma Attack
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FASTER
Record Dates: First submitted 2020-06-26; First posted 2020-11-05 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Asthma Attack; Asthma
MeSH Terms: conditions — Asthma | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Benralizumab (Experimental): Benralizumab 30 mg given in the form of subcutaneous injection every 4 weeks for the first three doses, then every 8 weeks subsequently up till Week 48.
  Interventions: Drug: Benralizumab 30 MG/ML [Fasenra]
- Placebo (Placebo Comparator): Normal Saline given subcutaneously every 4 weeks for the first three doses, then every 8 weeks subsequently up till Week 48.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Benralizumab 30 MG/ML [Fasenra] — Benralizumab/placebo initiated at an acute severe asthma exacerbation, then continued over a period of 48 weeks
  Other Names: Fasenra
  Arms: Benralizumab
Drug: Placebos — Benralizumab/placebo initiated at an acute severe asthma exacerbation, then continued over a period of 48 weeks
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Approximately 300 million people have asthma worldwide and 400,000 people died from asthma globally in 2015 (GINA Asthma). Singapore's asthma mortality and hospitalisation rates are several times higher than OECD countries. Spot Blood eosinophil count (BEC) during an acute exacerbation of asthma was a predictor of more severe respiratory failure and was associated with future acute health care utilization (HR 1.8, 95% CI 1.1-2.9, p=0.02) in a previous study conducted across 4 ICUs in Singapore. Benralizumab, an anti-IL5 receptor α monoclonal antibody causes rapid depletion of blood eosinophils and reduces asthma exacerbations when given over 12-month duration in patient with Severe Eosinophilic Asthma. However, the efficacy of Benralizumab when given during an acute exacerbation of asthma in reducing future exacerbations or severity of asthma exacerbation is relatively unexplored. A Phase 2A randomized double-blind placebo-controlled trial involving the use of one dose of the intravenous formulation of Benralizumab (0.3 mg/kg or 1.0mg/kg) in patients presenting with acute asthma exacerbation did not demonstrate difference in the proportion of subjects with >/=1 asthma exacerbation at 12 weeks when compared to placebo (33.3% vs. 38.9%; P=0.67). However, compared with placebo, Benralizumab reduced asthma exacerbation rates by 49% (3.59 vs 1.82; P=0.01) and exacerbations resulting in hospitalization by 60% (1.62 vs 0.65; P=.02) in the combined groups at 12 weeks (secondary outcomes).

Benralizumab, an anti-IL5 receptor α monoclonal antibody causes rapid depletion of blood eosinophils and reduces asthma exacerbations when given over 12-month duration in patient with Severe Eosinophilic Asthma.

This study aims to look at whether subcutaneous administration of Benralizumab when initiated during an acute severe asthma exacerbation and then continued over 48 weeks period can increase time to first exacerbation compared to placebo as well as other key secondary outcome such as hospital readmission and health care utilization.

We hypothesise that administration of Benralizumab when initiated during an acute severe asthma exacerbation and then continued over 48 weeks period can increase time to first exacerbation compared to placebo as well as other key secondary outcome such as hospital readmission and health care utilization.

DETAILED DESCRIPTION:
The efficacy of Benralizumab when given during an acute exacerbation of asthma in reducing future exacerbations or severity of asthma exacerbation is relatively unexplored. A Phase 2A randomized double-blind placebo-controlled trial involving the use of one dose of the intravenous formulation of Benralizumab (0.3 mg/kg or 1.0mg/kg) in patients presenting with acute asthma exacerbation did not demonstrate difference in the proportion of subjects with >/=1 asthma exacerbation at 12 weeks when compared to placebo (33.3% vs. 38.9%; P=0.67). However, compared with placebo, Benralizumab reduced asthma exacerbation rates by 49% (3.59 vs 1.82; P=0.01) and exacerbations resulting in hospitalization by 60% (1.62 vs 0.65; P=.02) in the combined groups at 12 weeks (secondary outcomes).

The purpose of this study is to look at whether Benralizumab, an anti-IL5 receptor α monoclonal antibody given subcutaneously compared to placebo given subcutaneously, can increase time to first exacerbation, reduce health care utilisation and improve other asthma outcomes in patients presenting with acute severe asthma exacerbation requiring hospitalisation. Randomized double-blind placebo-controlled trial design was chosen to reduce selection bias by randomisation and concealment of allocation, reduce analysis or interobserver ascertainment bias by blinding, and reduce bias introduced by exclusion after randomisation by using Intention- to-treat (ITT) analysis. In addition, biomarker stratified approach using spot BEC < or >/= 300 cells/microL during an acute exacerbation will be used to evaluate its role as a predictive biomarker for response to Benralizumab.

The study aims to recruit 128 patients over a 2-year period at Singapore General Hospital and Changi General Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with severe asthma exacerbation requiring hospital admission
* Subjects aged 21 to 65 years with a physician diagnosis of asthma for greater than or equal to 1 year
* Subjects with 2 or more exacerbations in the past 12 months
* On maintenance of medium to high dose ICS/LABA (GINA Step 4 and 5) for at least 6 months
* Blood Eosinophil count of ≥ 150 cells/microL at time of admission or ≥ 300 cells/microL documented over the past 52 weeks
* Informed consent obtained

Exclusion Criteria:

* Subjects with asthma exacerbations who are treated and then discharged from ED within 24 hours
* Subjects with a physician diagnosis of COPD, bronchiectasis
* Smokers > 20 pack years
* Anaphylactic/anaphylactoid reaction presenting with bronchospasm
* Other known causes of eosinophilia besides asthma (e.g. parasitic infection)
* Subjects who are deemed by investigators to have with life expectancy of < 12 months (any cause)
* Subjects who are already on investigational drug or has been participating in another clinical study with an investigational product during the last 6 months
* Female subjects who are pregnant or planning pregnancy. All subjects should refrain from family planning during and 4 months following the last dose. Male subjects should refrain from fathering a child or donating sperm during the study and 4 months following the last dose
* Subjects with known history of allergy or reaction to any component of the investigational product formation
* Subjects with history of primary immunodeficiency
* Subjects who have received Xolair (anti-IgE mAb) within 4 months before randomization
* Subjects who receive immunoglobulin or blood products within 30 days before randomization

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2021-06-02 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Time to first exacerbation in patients with a severe asthma exacerbation with raised blood eosinophil count | Change from baseline (Day 1) to 52 weeks
  Time to first exacerbation requiring either oral corticosteroid (OCS) use and/or an unscheduled visit to the Emergency Department or hospitalization

SECONDARY OUTCOMES:
Time to hospital readmission due to asthma exacerbation (Key Secondary outcome) | Baseline (Day 1) to 52 weeks
  Time to hospital readmission due to asthma exacerbation
Rate of severe exacerbation (i.e. requiring admission to hospital for asthma exacerbation) | Baseline (Day 1) to 52 weeks
  NUmber of severe exacerbation (i.e. requiring admission to hospital for asthma exacerbation)
Hospital LOS (index admission and subsequent admissions) | Change from baseline (Day 1) to 52 weeks
  Total hospital LOS
Need for Intensive Care Unit (ICU) admission with/without mechanical ventilation during the index admission | Baseline (Day 1) to index admission discharge date
  ICU admission during index admission
Hospital survival post admission (index admission) | Baseline (Day 1) to index admission discharge date
  Hospital survival for index admission
Total OCS burden | Baseline (Day 1) to 52 weeks
  Cumulative OCS dose
Total number of exacerbations requiring emergency healthcare utilization (including ED, polyclinic visits, Specialist outpatient visits) | Baseline (Day 1) to 52 weeks
  Total number of emergency healthcare utilization for exacerbations
Pre/post bronchodilator Forced Expiratory Volume 1s (FEV1), FVC, FEV1/FVC at baseline and at 52 weeks | Change from baseline (Day 1) to 52 weeks
  Change in Pre/post bronchodilator Forced Expiratory Volume 1s (FEV1), FVC, FEV1/FVC
Blood eosinophil counts (serial measurement over 52 weeks) | Change from baseline (Day 1) to 52 weeks
  Change in blood eosinophils
GINA assessment of symptom control | Change from baseline (Day 1) to 52 weeks
  Change in GINA assessment of symptom control ( Well controlled, Partly controlled or Uncontrolled)
Asthma Control Questionnaire 7 (ACQ 7) | Change from baseline (Day 1) to 52 weeks
  Change in Asthma Control Questionnaire 7 (ACQ 7) Scores range from 0-6( higher is worse). A score of 0.0-0.75 is classified as well-controlled asthma; 0.75-1.5 is a grey zone; and >1.5 is poorly controlled asthma. The minimum clinically important difference is 0.5
St George's Respiratory Questionnaire (SGRQ) | Change from baseline (Day 1) to 52 weeks
  Change in St George's Respiratory Questionnaire (SGRQ) The SGRQ total score is made up of 2 parts : Part 1 addresses the frequency of respiratory symptoms and Part 2 addresses the patient's current state. Data is entered into the calculator and scores will be generated ( 0 to 100). The lower the score, the better.

OTHER OUTCOMES:
Adverse Events | Change from baseline (Day 1) to 52 weeks
  To evaluate adverse events, serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Mariko Koh, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Foreign, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yii ACA, Tay TR, Puah SH, Lim HF, Li A, Lau P, Tan R, Neo LP, Chung KF, Koh MS. Blood eosinophil count correlates with severity of respiratory failure in life-threatening asthma and predicts risk of subsequent exacerbations. Clin Exp Allergy. 2019 Dec;49(12):1578-1586. doi: 10.1111/cea.13465. Epub 2019 Aug 6. PMID 31310686
- [Result] Nowak RM, Parker JM, Silverman RA, Rowe BH, Smithline H, Khan F, Fiening JP, Kim K, Molfino NA. A randomized trial of benralizumab, an antiinterleukin 5 receptor alpha monoclonal antibody, after acute asthma. Am J Emerg Med. 2015 Jan;33(1):14-20. doi: 10.1016/j.ajem.2014.09.036. Epub 2014 Oct 5. PMID 25445859
- [Result] Bleecker ER, FitzGerald JM, Chanez P, Papi A, Weinstein SF, Barker P, Sproule S, Gilmartin G, Aurivillius M, Werkstrom V, Goldman M; SIROCCO study investigators. Efficacy and safety of benralizumab for patients with severe asthma uncontrolled with high-dosage inhaled corticosteroids and long-acting beta2-agonists (SIROCCO): a randomised, multicentre, placebo-controlled phase 3 trial. Lancet. 2016 Oct 29;388(10056):2115-2127. doi: 10.1016/S0140-6736(16)31324-1. Epub 2016 Sep 5. PMID 27609408
- [Result] FitzGerald JM, Bleecker ER, Nair P, Korn S, Ohta K, Lommatzsch M, Ferguson GT, Busse WW, Barker P, Sproule S, Gilmartin G, Werkstrom V, Aurivillius M, Goldman M; CALIMA study investigators. Benralizumab, an anti-interleukin-5 receptor alpha monoclonal antibody, as add-on treatment for patients with severe, uncontrolled, eosinophilic asthma (CALIMA): a randomised, double-blind, placebo-controlled phase 3 trial. Lancet. 2016 Oct 29;388(10056):2128-2141. doi: 10.1016/S0140-6736(16)31322-8. Epub 2016 Sep 5. PMID 27609406